CLINICAL TRIAL: NCT05268029
Title: Making HD Voices Heard - A Pilot Study on the myHDstory™ Platform
Brief Title: Making HD Voices Heard
Status: Completed | Type: Observational
Sponsor: Huntington Study Group (Network)
Responsible Party: Sponsor
Other Study IDs: Making HD Voices Heard
Record Dates: First submitted 2021-12-27; First posted 2022-03-07 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Huntington Disease
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Pilot Study, Making HD Voices Heard, will ask people living with HD to report what they experience and how they function.

DETAILED DESCRIPTION:
The Huntington Study Group (HSG) myHDstory™ Platform is an online, observational research platform that will host the Pilot Study, Making HD Voices Heard. The Pilot Study will ask people living with HD to report what they experience and how they function. Participants will provide self-reported information using their own compatible smartphones, laptops, desktops, or tablets. Participants will be asked to reply to a series of questions, including open-ended questions that will be transcribed by voice (microphone voice-to-text transcription) or keyboard-entered text to record what they experience in their own words.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 years and older
* Willing and able to provide informed consent electronically.
* Individuals answering as a participant must self-report they have been diagnosed with HD by a doctor.
* Ability to answer online questions or direct someone else to enter answers for them.
* Ability to ambulate independently and take care of some of his or her personal needs.
* Ability to read and understand English.
* Willing to create a unique identifier based on personal demographic information.
* Residing in the United States or its territories
* Owning or having access to an electronic device and secure internet connectivity

Exclusion Criteria:

An individual who does not meet all the inclusion criteria will be excluded from participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals who have been diagnosed with Huntington disease.
Sampling Method: Non-Probability Sample
Enrollment: 698 (Actual)
Dates: Start 2022-03-23 (Actual); Primary Completion 2023-10-11 (Actual); Study Completion 2023-10-11 (Actual)

PRIMARY OUTCOMES:
The ability to successfully consent and enroll at least 200 HD participants who have early to mid-stage manifest HD. | 3 months
  Ability to successfully consent and enroll at least 200 manifest HD participants (independent or with help of assistants) within three months as measured by the number of help line calls or emails received requesting technical or clinical support.
Participants' ability to successfully complete online self-reported questionnaires. | 3 months
  Participants' ability to successfully complete online self-reported questionnaires as measured by the number of completed questionnaires.
Utility and informativeness of data collected. | 9 months
  Utility and informativeness of capturing, extracting, curating, and analyzing verbatim responses to open-ended questions in the form of the HD-Patient Report of Problems (HD-PROP).

CONTACTS AND LOCATIONS:
Overall Officials: Karen E Anderson, MD, Principal Investigator — Georgetown University
Locations (1):
- Huntington Study Group, Rochester, New York, United States